CLINICAL TRIAL: NCT06733129
Title: Best Hypnotic Drug Choice for Rapid Sequence Induction in the Operating Room: a 3-arm Randomized Trial
Brief Title: Best Hypnotic Drug Choice for Rapid Sequence Induction in the Operating Room
Acronym: HYPNOTIKS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC24_0389
Record Dates: First submitted 2024-12-02; First posted 2024-12-13 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Rapid Sequence Induction
Keywords: Rapid sequence induction; Full stomach patient; hypotension; propofol; ketamine; ketofol; general anesthesia
MeSH Terms: conditions — Hypotension | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- KETOFOL (Experimental): Ketofol: combination of Ketamine and Propofol : consecutive direct IV injection of Ketamine 1 mg/kg and Propofol 1 mg/kg after completing pre-oxygenation
  Interventions: Drug: combination of Ketamine and Propofol
- KETAMINE (Experimental): direct IV injection at dosage of 2 mg/kg after completing pre-oxygenation
  Interventions: Drug: direct IV injection
- PROPOFOL (Active Comparator): direct IV injection at dosage of 2 mg/kg after completing pre-oxygenation.
  Interventions: Drug: direct IV injection

INTERVENTIONS:
Drug: direct IV injection — direct IV injection at dosage of 2 mg/kg (adjusted body weight if BMI > 30) after completing pre-oxygenation
  Arms: KETAMINE; PROPOFOL
Drug: combination of Ketamine and Propofol — combination of Ketamine and Propofol described above: consecutive direct IV injection of Ketamine 1 mg/kg and Propofol 1 mg/kg (adjusted body weight if BMI > 30). Dilution are not necessary.
  Arms: KETOFOL

SUMMARY:
The best hypnotic choice to optimize the balance between good intubation condition quality and hemodynamic stability during RSI performed in the operating theatre remained to be investigated.

Therefore, a randomized study evaluating the efficacy of propofol, ketamine, and a combination of both is appropriate. So, we designed the HyPnotiKs randomized controlled study to investigate the efficacy of these hypnotic drugs in patients undergoing RSI in the operating theatre. The primary endpoint will be the successful tracheal intubation at the first attempt without major arterial hypotension event.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 - 80 years' old
* female* and male

  * ≥ 1 risk factor of aspiration of gastric contents defined as
  * preoperative fasting period of less than 6 hours,
  * occlusive syndrome, functional ileus, vomiting episode within the last 12 hours,
  * orthopaedic trauma within the last 12 hours,
  * medical history of symptomatic gastroesophageal reflux or hiatus, hernia or gastroparesis or dysautonomia or gastroesophageal surgery with sphincter dysfunction)
* patient requiring orotracheal intubation during general anaesthesia in the operating room.
* patient or his/her next of kin written informed consent or emergency procedure
* failure to discontinue GLP1 analogue as recommended (exenatide, liraglutide, albiglutide, taspoglutide, lixisenatide)

Exclusion Criteria:

* predicted impossible tracheal intubation (≥ 1 of the following criteria: patient with known intubation complications, Mallampati score IV, Thyromental Distance ≤ 4.0 cm, Mouth Opening < 3 cm, Sternomental Distance < 12.5 cm, significant modification of the airway due to congenital, cancer, trauma or burning lesions (non-exhaustive list)) [30]
* preoperative arterial hypotension (MAP < 65 mmHg or under catecholamine)
* preoperative respiratory distress syndrome (SpO2 < 90% in room air)
* contraindications to the use of ketamine and/or propofol and/or NMB:

  * allergy to the active substance or to one of the excipients or to soy or peanuts,
  * porphyria
  * intracranial hypertension
  * uncontrolled arterial hypertension (systolic arterial pressure > 180 mmHg)
  * personal or family history of known malignant hyperthermia, congenital muscular dystrophy, myasthenia, a known congenital deficit in plasma pseudocholinesterase
* pregnancy or breast-feeding woman
* patients under court protection or guardianship
* absence of insurance covering health costs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1218 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2027-04-14 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
proportion of patients with successful intubation at first attempt and without post-induction hypotension | within 10 minutes after the start of the hypnotic injection
  The main objective of the study is to compare the efficacies of ketamine alone and ketamine-propofol combination compared to standard doses of propofol to achieve successful tracheal intubation on the first attempt without hemodynamic hypotension in patients at risk of aspiration of gastric contents in the operating room. The composite primary outcome is the proportion of patients with successful intubation at first attempt and without post-induction hypotension defined by a mean arterial pressure ≤ 60 mmHg within 10 minutes after the start of the hypnotic injection.

SECONDARY OUTCOMES:
rates of arterial hypotension episodes | within 10 minutes after the start of the hypnotic injection
  rates of arterial hypotension episodes as defined in primary endpoint within 10 minutes after induction of anaesthesia compared between the three study groups
rates of tracheal intubation at the first attempt | within 10 minutes after the start of the hypnotic injection
  rates of tracheal intubation at the first attempt compared between the three study groups
quality of the intubation | within 10 minutes after the start of the hypnotic injection
  In the operating theatre (within 10 minutes after the start of the hypnotic injection): intubation difficulty scale (IDS-3) values
quality of the intubation | within 10 minutes after the start of the hypnotic injection
  In the operating theatre (within 10 minutes after the start of the hypnotic injection): Cormack-Lehane score values (from 1 to 4)
  * Cormack 1: The glottis is seen in its entirety
  * Cormack 2: Only the posterior half of the glottis is seen
  * Cormack 3: Only a small part of the glottis is seen
  * Cormack 4: The glottis is hidden by the epiglottis and tongue.
rates of vasopressor use and volume of intravenous fluids for vascular filling (from entry into the operating theatre to induction and from induction to recovery room) | within 10 minutes after the start of the hypnotic injection
  In the operating theatre (within 10 minutes after the start of the hypnotic injection): rates of vasopressor use and volume of intravenous fluids for vascular filling (from entry into the operating theatre to induction and from induction to recovery room)
volume of intravenous fluids for vascular filling | up to relapse of the recovery room (up to 7 days after surgery)
  volume of intravenous fluids for vascular filling (from entry into the operating theatre to induction and from induction to recovery room)
time between administration of hypnotic and tracheal intubation | within 10 minutes after the start of the hypnotic injection
  Efficacy of ketamine and / or ketamine-propofol combination compared to standard doses of propofol on the prevention of postoperative complications in the operating theatre (within 10 minutes after the start of the hypnotic injection) : - time between administration of hypnotic (start of anesthetic induction) and tracheal intubation (defined as the 6th capnography curve)
values of heart rate | within 10 minutes after the start of the hypnotic injection
  Efficacy of ketamine and / or ketamine-propofol combination compared to standard doses of propofol on the prevention of postoperative complications in the operating theatre (within 10 minutes after the start of the hypnotic injection) : values of heart rate measured every 1 minute from pre-oxygenation to 10 minutes after the start of the hypnotic injection
values of SpO2 | within 10 minutes after the start of the hypnotic injection
  Efficacy of ketamine and / or ketamine-propofol combination compared to standard doses of propofol on the prevention of postoperative complications in the operating theatre (within 10 minutes after the start of the hypnotic injection): SpO2 measured every 1 minute from pre-oxygenation to 10 minutes after the start of the hypnotic injection
values of blood pressure | within 10 minutes after the start of the hypnotic injection
  Efficacy of ketamine and / or ketamine-propofol combination compared to standard doses of propofol on the prevention of postoperative complications in the operating theatre (within 10 minutes after the start of the hypnotic injection): systolic/diastolic/mean blood pressure measured every 1 minute from pre-oxygenation to 10 minutes after the start of the hypnotic injection
rates of pulmonary aspiration of gastric contents | within 10 minutes after the start of the hypnotic injection
  Efficacy of ketamine and / or ketamine-propofol combination compared to standard doses of propofol on the prevention of postoperative complications in the operating theatre (within 10 minutes after the start of the hypnotic injection): rates of pulmonary aspiration of gastric contents during the intubation procedure
Tolerance of ketamine and / or ketamine-propofol combination compared to standard doses of propofol | during stay in the recovery room
  Tolerance of ketamine and / or ketamine-propofol combination compared to standard doses of propofol in the recovery room by postoperative Nu-DESC (Nursing Delirium Screening Scale) score value compared with preoperative score From 0 to 10
Tolerance of ketamine and / or ketamine-propofol combination compared to standard doses of propofol | during stay in the recovery room
  Tolerance of ketamine and / or ketamine-propofol combination compared to standard doses of propofol in the recovery room: need of sedative therapy in the recovery room to treat a delirium episode.
Tolerance of ketamine and / or ketamine-propofol combination compared to standard doses of propofol | during stay in the recovery room (up to 7 days after induction)
  Tolerance of ketamine and / or ketamine-propofol combination compared to standard doses of propofol in the recovery room: Use of ketamine and total dose during intervention and total dose of ketamine in recovery room.
Tolerance of ketamine and / or ketamine-propofol combination compared to standard doses of propofol | within 7 days after the start of the hypnotic injection
  Tolerance of ketamine and / or ketamine-propofol combination compared to standard doses of propofol in the recovery room:
  Up to day 7:
  * rates of major cardiovascular complications defined as: cardiac arrest, sustained arrhythmia, myocardial infarction, stroke (total, ischaemic, and haemorrhagic), coronary revascularization or admission to ICU for acute heart failure
  * rates of mortality at day 7

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - Chr Angers, Angers
  - CHRU de Brest Hôpital Cavale Blanche, Brest
  - Ch Louis Pasteur, Chartres
  - CHU Dijon, Dijon
  - CHU Grenoble Alpes, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - APHP Bicêtre, Le Kremlin-Bicêtre
  - CH Le Mans, Le Mans
  - CHU Lille Hopital Salengro, Lille
  - CHU Lille Hôpital Claude Huriez, Lille
  - CHU Lyon Hôpital Sud, Lyon
  - HCL Lyon Croix-Rousse, Lyon
  - Chu Nantes (Laennec), Nantes
  - Chu Nantes, Nantes
  - APHP St-Antoine, Paris
  - APHP Tenon, Paris
  - CHU Poitiers, Poitiers
  - Hopital Foch, Suresnes
  - CHU Toulouse Hôpital Purpan, Toulouse
  - CHU Toulouse Hôpital Rangueil, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grillot N, Volteau C, Quillet P, Ambrosi X, Caillard A, David JS, Blet A, Bouzat P, Blanchet L, Bruneau N, Chebbi N, Saint-Genis Q, Figueiredo S, Guinot PG, Joosten A, Le Guen M, Labaste F, Lasocki S, Oudot M, Pommier M, Rousseleau D, Verdonk F, Tching-Sin M, Faurel-Paul E, Counille F, Cosse C, Flattres Duchaussoy D, Cinotti R, Roquilly A. Best hypnotic drug choice for rapid sequence induction in the operating room: study protocol for a 3-arm superiority open-labeled randomized controlled trial with blinded evaluation of the primary outcome (the HyPnotiKs study). Trials. 2026 Jan 16. doi: 10.1186/s13063-026-09452-6. Online ahead of print. PMID 41546091